CLINICAL TRIAL: NCT03121001
Title: A Phase II Study of HLA-Haploidentical Stem Cell Transplantation to Treat Clinically Aggressive Sickle Cell Disease
Brief Title: Study of HLA-Haploidentical Stem Cell Transplantation to Treat Clinically Aggressive Sickle Cell Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Damiano Rondelli, MD, Professor, Hematology, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-1152
Record Dates: First submitted 2017-04-14; First posted 2017-04-19 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — thymoglobulin; fludarabine; Cyclophosphamide; Whole-Body Irradiation; Sirolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Subject treatment (Experimental): Patients will receive the following conditioning regimen: ATG, fludarabine (6 days before stem cell infusion), cyclophosphamide, and total body irradiation. The stem cell product will be infused according to BMT unit policy. Patients will also receive GVHD prophylaxis which will consist of cyclophosphamide, sirolimus, and mycophenolate mofetil according to the protocol. Post-transplant evaluation will be done as per standard care with study data collected at days 30, 60, 100, 180, 365, and annually thereafter.
  Interventions: Drug: ATG; Drug: fludarabine; Drug: cyclophosphamide; Radiation: Total body irradiation; Procedure: Stem cell infusion; Drug: Sirolimus; Drug: mycophenolate mofetil

INTERVENTIONS:
Drug: ATG — 0.5 mg/kg IV on day -9, and 2 mg/kg on days -8 and day -7
  Other Names: Thymoglobulin®
Drug: fludarabine — 30 mg/m2 IVPB daily for day -6 (6 days before stem cell infusion) through day -2
Drug: cyclophosphamide — 14.5 mg/kg IV on days -6 and -5 and 50 mg/kg/d on days +3 and +4
Radiation: Total body irradiation — 3 Gy on day -1
Procedure: Stem cell infusion — Stem cell product infused according to BMT unit policy on day 0.
Drug: Sirolimus — loading dose of 15 mg followed by 5 mg per day on day +5
Drug: mycophenolate mofetil — 1 g every 8 h (until day 35) will be started on day 5

SUMMARY:
The study is a Phase II clinical trial. Patients will receive intensity modulated total body irradiation (TBI) at a dose of 3 Gy with standard fludarabine/ i.v. cyclophosphamide conditioning prior to human leukocyte antigen (HLA)-haploidentical hematopoietic stem cell transplant (HSCT).

The primary objective of the study is to determine the engraftment at Day +60 following HLA-haploidentical hematopoietic stem cell transplant protocol using immunosuppressive agents and low-dose total body irradiation (TBI) for conditioning and post-transplant cyclophosphamide in patients with sickle cell disease.

ELIGIBILITY:
Patient Eligibility:

1. Patients with sickle cell disease are eligible if they have any of the following complications:

   1.1 Stroke or central nervous system event lasting longer than 24 hours 1.2 Frequent vaso-occlusive pain episodes, defined as ≥ 3 per year requiring emergency room, acute care center, hospital admissions, or home bedrest leading to absence from work or school. 1.3 Recurrent episodes of priapism, defined as ≥ 2 per year requiring emergency room visits 1.4 Acute chest syndrome with recurrent hospitalizations, defined as ≥ 2 lifetime events 1.5 Red-cell alloimmunization (≥ 2 antibodies) during long-term transfusion therapy 1.6 Bilateral proliferative retinopathy with major visual impairment in at least one eye 1.7 Osteonecrosis of 2 or more joints 1.8 Sickle cell nephropathy, defined by a GFR < 90mL/min/1.73m2 or the presence of macroalbuminuria (urine albumin > 300 mg/g creatinine) 1.9 Pulmonary hypertension, defined by a mean pulmonary arterypressure >25mmHg
2. Age 16-60 years
3. Karnofsky performance status of 60 or higher (Appendix A)
4. Adequate cardiac function, defined as left ventricular ejection fraction ≥ 40%
5. Adequate pulmonary function, defined as diffusion lung capacity of carbon monoxide ≥ 50% predicted (after adjustment for hemoglobin concentration)
6. Estimated GFR ≥ 50mL/min/1.73m2 as calculated by the modified MDRD equation
7. ALT ≤ 3x upper limit of normal
8. HIV-negative
9. Patient is not pregnant
10. Patient is able and willing to sign informed consent
11. Patient does not have a fully HLA-matched sibling donor
12. Patient has an HLA-haploidentical relative

Donor Eligibility Relatives (parents, offspring, siblings, aunts/uncles, cousins) will be tested by molecular typing of HLA class I (A, B, and C) and class II (DRB1) at low resolution. Only those that are an HLA-haploidentical match (≥ 4/8) will be considered as a potential donor. NOTE: If during testing, a fully HLA-matched sibling donor is found and is willing to donate his/her stem cells, the potential subject will not be eligible for this protocol.

Donor consent will be obtained as per standard protocol of the bone marrow transplant unit.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-03-20 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Estimate the number of patients who engraft by Day +60 | Up to Day +60
  Patients who achieve < 5% peripheral blood donor chimerism by Day +30 and do not have a Day +60 measure will be regarded as failing to achieve full donor chimerism by Day +60; patients who achieve > 5% donor chimerism by Day +30 but do not have a Day +60 measure will be considered nonevaluable for the primary endpoint.

SECONDARY OUTCOMES:
Disease free survival | Up to Day +60
  Using the Kaplan-Meier method, the probability of EFS will be estimated and reported with 90% confidence intervals. The proportion of patients who are alive will also be estimated with a 90% exact binomial confidence interval. Cumulative incidences of transplant related mortality will be estimated separately using Grey's method.
Overall survival | Up to Day +60
  Using the Kaplan-Meier method, the probability of overall survival will be estimated and reported with 90% confidence intervals. The proportion of patients who are alive will also be estimated with a 90% exact binomial confidence interval. Cumulative incidences of transplant related mortality will be estimated separately using Grey's method.
Adverse Effects | Up to Day +60
  The cumulative incidence of acute (grade II-IV, grade III-IV) and chronic GVHD will be estimated through competing-risk analysis using Grey's method, wherein graft failure, and death are competing risks for GVHD. Other selected toxicities (including rates of infection) will be reported descriptively.

CONTACTS AND LOCATIONS:
Overall Officials: Damiano Rondelli, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States